CLINICAL TRIAL: NCT04905342
Title: An Open-label, Randomized, Evaluate the Pharmacokinetics and the Safety of NVP-1805 Compared to Coadministration of NVP-1805-R1 With NVP-1805-R2 in Healthy Adult Volunteers
Brief Title: NVP-1805 Compared to Coadministration of NVP-1805-R1 With NVP-1805-R2 in Healthy Adult Volunteers
Acronym: BE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NVP Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NVP-1805_BE-02
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: single-dose, crossover study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NVP-1805 (Experimental): NVP-1805 (80/10/20.8mg)
  Interventions: Drug: NVP-1805
- NVP-1805-R1 and NVP-1805-R2 (Active Comparator): coadministration of NVP-1805-R1(80mg) and NVP-1805-R2(10/20.8mg)
  Interventions: Drug: NVP-1805-R1and NVP-1805-R2

INTERVENTIONS:
Drug: NVP-1805 — orally, once daily on Period 1 and Period 3 (or Period 2 and Period 4) (NVP-1805 80/10/20.8mg)
  Arms: NVP-1805
Drug: NVP-1805-R1and NVP-1805-R2 — orally, once daily on Period 1 or Period 3 (or Period 2 and Period 4) (NVP-1805-R1 80mg, NVP-1805-R2 10/20.8mg)
  Arms: NVP-1805-R1 and NVP-1805-R2

SUMMARY:
The purpose of this study is to compare the pharmacokinetics of NVP-1805 and coadministration of NVP-1805-R1 with NVP-1805-R2.

DETAILED DESCRIPTION:
Evaluate pharmacokinetics and safety of NVP-1805 compared to coadministration of NVP-1805-R1 with NVP-1805-R2

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult subjects who signed informed consent
* BMI of >18.0 kg/㎡ and <30.0 kg/㎡ subject, weight more than 50kg(45 kg or more for woman)

Exclusion Criteria:

* Subjects participated in another clinical trial within 6 months prior to administration of the study drug
* Inadequate subject for the clinical trial by the investigator's decision
* Subjects participated in another clinical trial within 6 months prior to administration of the study drug

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-08-14 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2022-01-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of plasma: AUClast | 0hours - 72hours
  period 1,2,3,4
Pharmacokinetics of plasma: Cmax | 0hours - 72hours
  period 1,2,3,4

CONTACTS AND LOCATIONS:
Overall Officials: Jaewoo Kim, M.D., Principal Investigator — H Plus Yangji Hospital
Locations (1):
- H Plus Yangji Hospital, Seoul, Nambusunhwan-ro, South Korea